CLINICAL TRIAL: NCT07028645
Title: Is Uroflowmetry Useful in Assessing Response to Pharmacological Treatment in Enuresis
Brief Title: Uroflowmetry and Nocturnal Enuresis
Status: Active, not recruiting | Type: Observational
Sponsor: Furkan Adem Canbaz (Other)
Responsible Party: Sponsor-Investigator, Furkan Adem Canbaz, Medical doctor, Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Organization: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Other Study IDs: Ivstrh - UF PMNE
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Enuresis, Nocturnal
Keywords: Uroflowmetry; Enuresis
MeSH Terms: conditions — Nocturnal Enuresis; Enuresis | interventions — Freezing; propiverine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Desmopressin 120mcg: Patients treated with desmopressin 120 mcg
  Interventions: Drug: desmopressin melt form 120 μg
- Desmopressin 240 mcg: Patients treated with desmopressin 240mcg
  Interventions: Drug: Desmopressin lyophilisate (Melt)
- Desmopressin 240 mcg + anticholinergic: Patients treated with desmopressin 240mcg + anticholinergic agent
  Interventions: Drug: Propiverine tablet

INTERVENTIONS:
Drug: desmopressin melt form 120 μg — Desmopressin 120 mcg will be used frist-line drug in the treatment of enuresis.
  Groups: Desmopressin 120mcg
Drug: Desmopressin lyophilisate (Melt) — Desmopressin 240 mcg will be used for the patients who have not responsive to desmopressin 120 mcg.
  Groups: Desmopressin 240 mcg
Drug: Propiverine tablet — Propiverine (a dose of 0.8 mg/ kg) will be used for the patients who have -response to treatment with desmopressin 240 mcg
  Groups: Desmopressin 240 mcg + anticholinergic

SUMMARY:
This study will evaluate the uroflowmetry parameters of patients which were treated for enuresis.

DETAILED DESCRIPTION:
A total of approximately 100 patients with enuresis will be evaluated retrospectively. Uroflowmetry parameters of these patients will be evaluated. For this purpose, patients will be divided to mainly three groups according to the treatment choices.

ELIGIBILITY:
Inclusion Criteria:

* Presence of enuresis nocturna
* Patients who have uroflowmetry test

Exclusion Criteria:

* Presence of lower urinary tract symptoms
* Presence of anatomical or neurological problems
* Patients with missing data

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who were treated for enuresis in pediatric urology clinic of Sancaktepe Sehit Prof Dr Ilhan Varank Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of days without bedwetting | 1 month
  Achievement of bedwetting in one or less night of a month

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Sehit Prof dr Ilhan Varank Training and Research Hospital, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kang BJ, Chung JM, Lee SD. Evaluation of Functional Bladder Capacity in Children with Nocturnal Enuresis According to Type and Treatment Outcome. Res Rep Urol. 2020 Sep 15;12:383-389. doi: 10.2147/RRU.S267417. eCollection 2020. PMID 32984086